CLINICAL TRIAL: NCT04788368
Title: TRECA - TREatment of Colorectal Adenomas and Early Colorectal CAncer in Region Västra Götaland
Acronym: TRECA
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: TRECA
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients treated with TEM - transanala microsurgery: Early rectal cancer treated with TEM - full thickness resection
  Interventions: Procedure: Surgical resection
- Patients treated with ESD: Early rectal cancer treated with the endoscopic treatment ESD - endoscopic submucosal resection
  Interventions: Procedure: Surgical resection
- Patients treated with EMR: Early rectal cancer treated with the endoscopic treatment EMR - endoscopic mucosal resection
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection with either of the above mentioned techniques

SUMMARY:
All early colorectal cancers (T1-T2) treated in the Region Västra Götaland from 2007-2020 will be evaluated. To establish the extent to which early colorectal cancers have been treated with local excision? How have treatment strategies changed over time? The study will provide information on where these patients have been treated in the Region Västra Götaland. During the study period, ESD was introduced as a treatment modality, and it will investigated how this may have influenced treatment strategies for complex adenomas. Clinical outcome measures will include recurrence rates and re-intervention rates for the respective treatments. Possible areas of improvement will be identified and determine if evidence based and best practice guidelines are met with the current treatment strategies in Region Västra Götaland.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer resected by local resection

Exclusion Criteria:

* All other types of resection or treatment for rectal cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rectal cancer treated with a local resection
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pathological clear margins | 1-2 months after surgery
  Pathological examination of the specimen showing free margins
Complications after surgery | 90 days after surgery
  Complications graded using the Clavien Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No